CLINICAL TRIAL: NCT05138068
Title: Social Anxiety MDMA-Assisted Therapy Investigation (SAMATI): A Randomized, Delayed Treatment Control Phase 2 Study of the Safety and Effectiveness of Manualized MDMA-Assisted Therapy for the Treatment of Social Anxiety Disorder
Brief Title: Social Anxiety MDMA-Assisted Therapy Investigation
Acronym: SAMATI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason B Luoma (Other)
Collaborators: Oregon Research Institute Center for Evaluation Services (Unknown); Multidisciplinary Association for Psychedelic Studies (Other); Portland Psychotherapy Clinic, Research, and Training Center (Other)
Responsible Party: Sponsor-Investigator, Jason B Luoma, CEO, Portland Psychotherapy Clinic, Research, and Training Center
Organization: Portland Psychotherapy Clinic, Research, and Training Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUSA5
Record Dates: First submitted 2021-11-15; First posted 2021-11-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Social Anxiety Disorder
Keywords: 3,4-methylenedioxymethamphetamine; MDMA; Psychotherapy; Mental Disorders; Hallucinogens; Serotonin Agents; Neurotransmitter Agents; Adrenergic Uptake Inhibitors; Adrenergic Agents; Neurotransmitter Uptake Inhibitors; Psychotropic Drugs; Anxiety disorders; Phobia, Social
MeSH Terms: conditions — Phobia, Social; Mental Disorders; Anxiety Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label delayed treatment study to assess the safety and effect of MDMA-assisted therapy in treating 20 participants diagnosed with moderate-to-severe social anxiety disorder (SAD) of the generalized subtype.
Masking Description: Primary outcome measures will be administered by blinded, independent raters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MDMA-assisted psychotherapy (Experimental): Two sessions of manualized MDMA-assisted psychotherapy with flexible dose of MDMA from 80 to 120 mg and optional supplemental dose 1.5 to 2 hours later. MDMA sessions are preceded by 3 non-drug preparatory psychotherapy sessions and followed by 3 integrative non-drug psychotherapy sessions.
  Interventions: Drug: MDMA; Behavioral: Psychotherapy
- Delayed treatment (Other): Participants randomly assigned to the delayed treatment control condition will wait 16 weeks and then receive MDMA-assisted therapy protocol described in the experimental arm of the study.
  Interventions: Drug: MDMA; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: MDMA — Two 8-hour experimental sessions will occur within the 11-session intervention in which participants will take a dose of MDMA. In the first Experimental Session, the initial dose will be 80 mg MDMA, with a supplemental dose of 40 mg 1.5 to 2 hours later unless contraindicated. In the second Experimental Session, the initial dose may be increased to 120 mg MDMA unless contraindicated with an additional dose of 40 mg 1.5 to 2 hours after the initial dose is given unless contraindicated.
  Other Names: 3,4-Methylenedioxymethamphetamine
Behavioral: Psychotherapy — Adjunctive, manualized psychotherapy will be provided by a team of two therapists during the MDMA-assisted therapy sessions

SUMMARY:
This is a randomized, open-label delayed treatment study to assess the safety and effect of MDMA-assisted therapy in treating 20 participants diagnosed with moderate-to-severe social anxiety disorder (SAD) of the generalized subtype. This study will obtain an estimate of effect size for two experimental sessions of MDMA-assisted therapy for the treatment of social anxiety disorder on measures of safety, social anxiety, functional outcomes, psychiatric symptoms, and putative mechanisms of action. The primary outcome for this study will be the Liebowitz Social Anxiety Scale (LSAS) administered by a blinded Independent Rater (IR). Other assessments, including physiological, self-report, and behavioral tasks will be used to assess other exploratory variables. An additional aim of the trial will be the development of a treatment manual for MDMA-AT for SAD for future research.

DETAILED DESCRIPTION:
SAD is a prevalent and disabling disorder characterized by intense fear of being scrutinized or negatively evaluated by others in social situations. SAD is the fourth most commonly diagnosed psychological disorder in the United States with onset commonly occurring in adolescence and assuming a chronic course even when treated. Evidence-based treatments for SAD exist, including medications and therapy, but a significant proportion of patients fail to improve, indicating the need for novel effective treatments.

3,4-methylenedioxymethamphetamine (MDMA) is a monoamine releaser and re-uptake inhibitor with indirect effects on neurohormone release. The combined neurobiological effects appear to reduce defenses and fear of emotional injury, enhance communication and introspection, and can increase empathy and compassion. MDMA may also enhance fear extinction learning in humans. The subjective effects of MDMA appear to create a productive psychological state that enhances the therapeutic process. These subjective effects of MDMA create a productive psychological state that enhances the therapeutic process for the treatment of SAD and other anxiety disorders. A Phase 2 MDMA-assisted therapy (MDMA-AT) trial sponsored by MAPS has provided preliminary evidence that social anxiety among adults with autism is treatable with two MDMA-AT sessions and associated non-drug preparatory and integrative psychotherapy (Danforth et al., 2018).

In this open-label Phase 2 study intended to gather supportive data on the safety and effectiveness of MDMA-assisted therapy (MDMA-AT), each of the 20 subjects will participate in two experimental sessions, with half proceeding immediately into treatment once enrolled, and half receiving the experimental treatment after an initial 16 week wait. This study involves a dose of MDMA administered during the Treatment Period with manualized therapy in two monthly Experimental Sessions. This 8-week Treatment Period is preceded by three 90-minute non-drug Preparatory Sessions. Each experimental Session is followed by three 90-minute non-drug Integrative Sessions of non-drug psychotherapy. The Primary Outcome measure is assessed by a blinded Independent Rater at study enrollment, at the primary outcome assessment point (2-weeks after the final integration session), and follow up assessment 26 weeks later. Participants will also be offered the chance to sign up for a long-term follow up extension study at the follow up assessments (with long-term follow up conducted 24 months post-treatment).

ELIGIBILITY:
Inclusion:

1. Are between the ages of 18 and 65 years old.
2. Live in the Portland, OR area.
3. Are fluent in speaking and reading English.
4. Are able to swallow pills.
5. Agree to have study visits recorded, including Experimental Sessions, assessments, and non-drug psychotherapy sessions.
6. Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
7. Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
8. If able to become pregnant, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
9. Agree to the necessary lifestyle modifications.
10. Able to identify support person who can stay with participant overnight after experimental sessions.
11. Suitable home environments to allow completion of all study procedures, including sufficient privacy and access to computer or mobile device with internet access.
12. At Screening, meet DSM-5 criteria for current SAD, generalized subtype.
13. At Screening, may have well-controlled hypertension that has been successfully treated with anti-hypertensive medicines, if they pass additional screening to rule out underlying cardiovascular disease.
14. At Screening, may have asymptomatic hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
15. At Enrollment confirmation for those in delayed treatment group, continue to meet criteria for SAD, generalized subtype.
16. Enrollment is allowed with glaucoma only with the approval of their ophthalmologist.

Exclusion:

1. Are not able to give adequate informed consent.
2. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of SAD or any other psychiatric disorder.
3. Are likely, in the investigator's opinion and via observation during the Preparatory Period, to lack social support or lack a stable living situation or supportive family/network.
4. Have any current problem which, in the opinion of the investigator or Study Physician, might interfere with participation.
5. Would present a serious risk to others as assessed by investigator, Study Physician, or study team.
6. Require certain excluded medications.
7. Have evidence or history of significant (controlled or uncontrolled) hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, or any other medical disorder judged by the investigator to significantly increase the risk of MDMA administration (participants with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded).
8. Have uncontrolled hypertension using the standard criteria of the American Heart Association (values of 140/90 millimeters of Mercury [mmHg] or higher assessed on three separate occasions).
9. Have a marked baseline prolongation of QT/QTc interval.
10. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
11. Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions.
12. Have symptomatic liver disease.
13. Have history of hyponatremia or hyperthermia.
14. Weigh less than 48 kilograms (kg).
15. Are pregnant, nursing, or are able to become pregnant and are not practicing an effective means of birth control.

Some eligibility criteria have been omitted to protect the integrity of the recruitment process. Full exclusion/inclusion criteria will be reported with results when recruitment is complete. In the interim, please contact research team to inquire about full inclusion/exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of MDMA-assisted therapy on severity of social anxiety disorder symptoms, as measured by total score on the Liebowitz Social Anxiety Scale (L-SAS). | Baseline, Primary outcome (2 weeks after final integration session), follow up (26-weeks after primary outcome)
  Primary outcome analyses are intent-to-treat comparing mean scores on the Liebowitz Social Anxiety Scale (LSAS) at post-treatment assessment point in the immediate treatment condition compared to the 16 week assessment in the delayed treatment condition. A participant is considered eligible for the ITT analysis if they have completed at least one Experimental Session and at least one LSAS assessment beyond baseline.
  The LSAS (Heimberg et al., 1999) is a 24-item, semi-structured interview on the severity of social anxiety disorder, which assesses fear (0 to 3 = none, mild, moderate, severe) and avoidance (0 to 3 = never, occasionally, often, usually) of 24 social situations over the previous week, providing an overall social anxiety severity rating and subscale scores for performance fear, performance avoidance, social fear, and social avoidance. Scores range from a minimum of 0 to maximum of 144 with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Evaluate the effectiveness of MDMA-assisted therapy for SAD in clinician-rated functional impairment, as measured by the mean change in item scores on the Sheehan Disability Scale (SDS). | Baseline, Primary outcome (2 weeks after final integration session), follow up (26 weeks after primary outcome)
  The SDS is a clinician-rated assessment of functional impairment (Sheehan, 1986). The items indicate degree of impairment in the domains of work/school, social life, and home life, with response options based on an eleven-point scale (0=not at all to 10=extremely), and five verbal tags (not at all, mildly, moderately, markedly, extremely) and has been validated for use in clinical trials (K. H. Sheehan & Sheehan, 2008). Higher scores indicate a higher degree of functional impairment.
Evaluate change in internalized shame as a potential process of change in MDMA-Assisted Therapy for SAD, as measured by mean change in Internalized Shame Scale (ISS) scores from pre- to post-treatment. | Baseline, Primary outcome (2 weeks after final integration session)
  The ISS is a 24-item self-report questionnaire measuring internalized shame that has been used in numerous studies of trait shame and has been demonstrated to have good construct validity and reliability in both clinical and nonclinical populations (del Rosario & White, 2006). Scores range from 0 - 96, with higher scores indicate higher levels of internalized shame.
Evaluate change in acceptance of self-conscious emotions as a potential process of change in MDMA-Assisted Therapy for SAD, as measured by mean change in Acceptance of Shame and Embarrassment Scale (ASES) scores from pre- to post-treatment. | Baseline, Primary outcome (2 weeks after final integration session)
  The ASES is a 17 item self-report measure (Sedighimornani, Rimes, Verplanken, & Gauntlett-Gilbert, 2019) intended to assess avoidance of shame and embarrassment, two emotions hypothesized to be central to the experience of SAD. The measure shows good internal reliability, factor structure, and correlation with theoretically meaningful constructs (Sedighimornani et al., 2019). Scores range from a minimum of 0 to maximum of 102 with higher scores indicating a better outcome.
Evaluate change in subjective belonging as a potential process of change in MDMA-Assisted Therapy for SAD, as measured by mean change in Interpersonal Needs Questionnaire (INQ) - Thwarted Belongingness scores from pre- to post-treatment. | Baseline, Primary outcome (2 weeks after final integration session)
  The 9-item Thwarted Belongingness subscale from the INQ (Freedenthal, Lamis, Osman, Kahlo, & Gutierrez, 2011) will be used to assess the degree to which participants feel a sense of belonging, connection, and closeness with others. Scores range from a minimum of 9 to maximum of 63 with higher scores indicating a worse outcome.
Evaluate change in self-concealment as a potential process of change in MDMA-Assisted Therapy for SAD, as measured by mean change in Hidden Self Scale (HSS) scores from pre- to post-treatment. | Baseline, Primary outcome (2 weeks after final integration session)
  The HSS (Levinson, Rodebaugh, Lim, & Fernandez, 2015) is a 4-item subscale of the Core Extrusion Schema-Revised and is thought to measure attempts to hide ones "true self" from others so as to avoid potential ostracism and rejection. This measure was created for use in SAD populations. The measure has demonstrated good psychometrics and the HSS subscale predicts the intensity of social interaction anxiety. Scores range from a minimum of 0 to maximum of 36 with higher scores indicating a worse outcome.
Evaluate change in self-compassion as a potential process of change in MDMA-Assisted Therapy for SAD, as measured by mean change in Self-Compassion Scale scores from pre- to post-treatment. | Baseline, Primary outcome (2 weeks after final integration session)
  The SCS short form (Raes, Pommier, Neff, & Van Gucht, 2010) is a 12-item self-report measure of self-compassion, or responding to one's own failure, suffering or inadequacies with kindness and compassion and recognizing one's own flaws and suffering as part of common human experience. The measure was modified in this study to assess self-compassion in the past week. Scores range from a minimum of 12 to maximum of 60 with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Luoma, Ph.D., Principal Investigator — Portland Psychotherapy Clinic, Research, and Training Center
Locations (1):
- Portland Psychotherapy Clinic, Research, & Training Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized data underlying publications as data sets accessible to other researchers. Requests for other data by outside researchers will be considered on a case-by-case basis.
Supporting Information: SAP, Analytic Code
Time Frame: At time of study publications
Access Criteria: Contact the sponsor-investigator to access data that is not publicly shared. Some deidentified data sets with be publicly shared.

REFERENCES:
- [Background] Danforth AL, Grob CS, Struble C, Feduccia AA, Walker N, Jerome L, Yazar-Klosinski B, Emerson A. Reduction in social anxiety after MDMA-assisted psychotherapy with autistic adults: a randomized, double-blind, placebo-controlled pilot study. Psychopharmacology (Berl). 2018 Nov;235(11):3137-3148. doi: 10.1007/s00213-018-5010-9. Epub 2018 Sep 8. PMID 30196397
- [Background] Luoma J, Lear MK. MDMA-Assisted Therapy as a Means to Alter Affective, Cognitive, Behavioral, and Neurological Systems Underlying Social Dysfunction in Social Anxiety Disorder. Front Psychiatry. 2021 Sep 27;12:733893. doi: 10.3389/fpsyt.2021.733893. eCollection 2021. PMID 34646176
- [Background] Luoma JB, Shahar B, Kati Lear M, Pilecki B, Wagner A. Potential processes of change in MDMA-Assisted therapy for social anxiety disorder: Enhanced memory reconsolidation, self-transcendence, and therapeutic relationships. Hum Psychopharmacol. 2022 May;37(3):e2824. doi: 10.1002/hup.2824. Epub 2021 Nov 5. PMID 34739165
- [Background] Danforth AL, Struble CM, Yazar-Klosinski B, Grob CS. MDMA-assisted therapy: A new treatment model for social anxiety in autistic adults. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Jan 4;64:237-49. doi: 10.1016/j.pnpbp.2015.03.011. Epub 2015 Mar 25. PMID 25818246
- [Derived] Lear MK, Smith SM, Pilecki B, Stauffer CS, Luoma JB. Social anxiety and MDMA-assisted therapy investigation: a novel clinical trial protocol. Front Psychiatry. 2023 Jul 14;14:1083354. doi: 10.3389/fpsyt.2023.1083354. eCollection 2023. PMID 37520237

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT05138068/SAP_000.pdf